CLINICAL TRIAL: NCT00670839
Title: Open-label, Randomized, and Multicenter Phase III Clinical Trial Comparing Immunogenicity of Double-dose (40 µg at S0, S4 and S24), Versus Standard Dose Vaccination (20 µg at S0, S4 and S24), Against Hepatitis B Virus in HIV-1-infected Patients Without Any Previous Immune Response After Primary Immunization Plus One Single Boost
Brief Title: Trial Comparing Two Strategies of Vaccination Against Hepatitis B in HIV-infected Patients Non Responding to Primary Immunization (B-BOOST)
Acronym: B-BOOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-005023-15; ANRS HB04 B-BOOST
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis B; HIV Infection
Keywords: Hepatitis B vaccination; GenHevac-B Pasteur; HIV infection
MeSH Terms: conditions — Hepatitis B; HIV Infections | interventions — GenHevac B Pasteur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): GenHevac-B 20 microgram intramuscular use at M0, M1 and M6
  Interventions: Biological: GenHevac-B
- B (Experimental): GenHevac-B 40 microgram intramuscular use at M0, M1 and M6
  Interventions: Biological: GenHevac-B

INTERVENTIONS:
Biological: GenHevac-B — 1 intramuscular injection of Genhevac-B® 20μg on day zero, month 1,and month 6
  Other Names: Sanofi Pasteur MSD
  Arms: A
Biological: GenHevac-B — 2 intramuscular injections of Genhevac-B® 20μg on day zero, month 1,and month 6
  Other Names: Sanofi Pasteur MSD
  Arms: B

SUMMARY:
HIV infected patients exposed to Hepatitis B virus are more susceptible to develop a chronic and severe liver disease, with a major risk of cirrhosis and liver cancer.

However, immune response to standard Hepatitis B vaccination is decreased in HIV-infected patients, compared to non HIV-infected individuals, and, in case of response, its durability has to be carefully followed up. This study compares the efficacy of two strategies of revaccination in HIV-infected patients who didn't respond to previous hepatitis B vaccination. Failure is defined by two conditions: non response to the primary immunization (2 to 4 single-dose injections received before the screening visit) and failure to a single 20 µg boost before being included in the study.

DETAILED DESCRIPTION:
Comparison of 2 revaccination strategies in randomized HIV-infected patients with T CD4 cell count above 200/mm3

Intervention:

1. Arm A: GenHevac-B® 20μg IM at M0, M1, M6
2. Arm B: GenHevac-B® 40μg IM at M0, M1, M6

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* T CD4 cell count number above 200 /mm3
* History of 2 to 4 injections of Hepatitis B vaccine, at any time in the past
* No history of Hepatitis B vaccination with a double-dose schedule
* No response to Hepatitis B vaccination: serology Hepatitis B negative (AgHBs, AbHBs and AbHBc negative) the previous twelve months and at the screening visit
* AbHBs titers below 10 IU/ml four weeks after the boost of Genhevac-B® 20μg preceding the randomization
* unchanged ARV treatment for the last 2 months for patients who are receiving ARV at the screening visit
* Undetectable HIV RNA for the last 6 months and on-going ARV for any patients with T CD4 cell level below 350/mm3
* HIV-1 plasma load below 100 000 copies per ml for patients without ARV
* Negative pregnancy test at the screening visit, and immediately before the Genhevac-B® 20 µg boost injection preceding the randomization

Exclusion Criteria:

* Acute cytolysis in the last 3 months with transaminases equal or above 5 times the upper limit of normal for HIV-HCV coinfected patients, or transaminases equal or above 2 times the upper limit of normal for non coinfected patients
* Any vaccine received during the month preceding the inclusion
* History of hypersensitivity to any component of GenHevac-B
* acute opportunistic infection treated the month before the screening visit
* Severe and acute pyretic infection or unexplained fever the week before inclusion
* Hemopathy or solid-organ cancer
* Prothrombin factor equal or below 50% and/or platelets equal or below 50 000 per mm3
* Immunosuppressive treatment or general corticotherapy (equal or above 0,5 mg per kg per day during at least 7 days) in the last 6 months before the screening visit
* Immunomodulating treatment (interferon, interleukine-2,…) in the last 6 months before the screening visit
* Splenectomy
* Decompensated cirrhosis (Child Pugh B or C)
* Renal failure (creatinine clearance below 50 ml/mn)
* Other severe immunocompromised condition not related to HIV infection (solid-organ transplantation, chemotherapy in the last 6 months,….)
* Any participation to another clinical trial plan until Week 28

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
rate of HIV-infected patients who seroconvert one month after the last vaccination. Seroconversion is defined as anti-HBs titers equal or above 10 mUI per ml | one month after the last vaccination (week 28)

SECONDARY OUTCOMES:
According to the vaccine strategy (single-dose or double-dose), comparison of AbHBs titers, permanence of humoral response, intensity of clinical and biological events, and predicting factors related to seroconversion | one month after the last injection ( week 28) and month 18
immunological substudy: to understand genetic link between some alleles of HLA-DR and non-response to immunization | at D0

CONTACTS AND LOCATIONS:
Overall Officials: David Rey, MD, Principal Investigator — Hôpital civil, Strasbourg, France; Fabrice Carrat, MD, Study Chair — Inserm U707 Paris France
Locations (1):
- Centre de Soins de l'Infection par le VIH NHC, Hôpitaux Universitaires Strasbourg, 1 place de l'hôpital, Strasbourg, France

REFERENCES:
- [Derived] Rey D, Piroth L, Wendling MJ, Miailhes P, Michel ML, Dufour C, Haour G, Sogni P, Rohel A, Ajana F, Billaud E, Molina JM, Launay O, Carrat F; ANRS HB04 B-BOOST study group. Safety and immunogenicity of double-dose versus standard-dose hepatitis B revaccination in non-responding adults with HIV-1 (ANRS HB04 B-BOOST): a multicentre, open-label, randomised controlled trial. Lancet Infect Dis. 2015 Nov;15(11):1283-91. doi: 10.1016/S1473-3099(15)00220-0. Epub 2015 Aug 6. PMID 26257021
- See also: Related Info — http://www.anrs.fr